CLINICAL TRIAL: NCT01611168
Title: Redesigning Medication Intensification Effectiveness Study for Diabetes
Brief Title: REMEDIES4D: REdesigning MEDication Intensification Effectiveness Study for Diabetes
Acronym: Remedies4D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO08040023
Record Dates: First submitted 2012-05-15; First posted 2012-06-04 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention)
- Intervention Group, treatment algorithms (Experimental)
  Interventions: Other: Treatment Algorithms

INTERVENTIONS:
Other: Treatment Algorithms — subjects in the intervention group will receive diabetes care from a well-trained registered nurse (RN) who will follow approved treatment algorithms/protocols for glycemia, high blood pressure, lipids and microalbuminuria.
  Arms: Intervention Group, treatment algorithms

SUMMARY:
The proposed research study aims to determine whether applying the University of Pittsburgh Medical Center Nurse-Directed Diabetes Management Protocols (NDMPs) leads to improved clinical outcome and process measures as recommended by American Diabetes Association (ADA), quality of life, treatment satisfaction and medication adherence for adults with diabetes, and favorable providers' satisfaction as compared to usual diabetes care. Furthermore, the cost-effectiveness of performing the NDMPs compared to usual diabetes care in primary care settings will also be assessed.

DETAILED DESCRIPTION:
This proposed study is a multi-practice, cluster-design, prospective randomized controlled trial with a total study intervention period of 12 months. This prospective randomized controlled trial will assess the effectiveness of performing NDMPs by the registered nurse supervised by a physician (the intervention group) in comparison with usual diabetes care (the usual care group) for adults with diabetes in primary care settings. The study population will be recruited from University of Pittsburgh Medical Center Community Medicine Inc. (CMI) primary care practices in urban and suburban communities surrounding Pittsburgh, PA. Among these CMI practices, ten practices receive diabetes education services from University of Pittsburgh Diabetes Institute and will be the intervention group. These diabetes education services will be enhanced by the addition of NDMPs intervention. In addition, we will select another 10 CMI practices to be the usual care group. This group receives standard diabetes education with no use of NDMPs. One-hundred and fifty participants will be recruited across practices within each study group (i.e., 300 in total). Outcomes assessed in this study include clinical outcome and process measures as recommended by ADA, participants' quality of life, treatment satisfaction, and medication adherence, and providers' satisfaction, and costs/expenditure. Assessments will be done at baseline, and three and 12 months after the study entry. Analysis of the study outcomes will be based on intention-to-treat to determine (1) within-group differences between the baseline and follow-up visits, and (2) between-group differences between the intervention group and the usual care group.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or greater
2. The diagnosis of type 2 diabetes of the subjects should be 1 year or more prior to the inception of this study
3. Subjects will be on medication treatment for their type 2 diabetes
4. Subjects' A1C levels should be higher than 7% for study entry
5. LDLc>100mg/d*l or
6. Blood Pressure >130/80*mg/dl
7. Any combination of the #4, 5 &6 At least one visit to the practice within the previous 12 months.

Exclusion Criteria:

1. Non-ambulatory
2. Gestational diabetes
3. Pregnant women (by self-report)
4. Subjects have received diabetes education services performed by the registered nurse from UPDI
5. Subjects are treated with exercise and diet only
6. Subjects are participating or will participate in other research studies
7. Subjects do not have insurance or cannot afford payments for diabetes care/treatment
8. Subjects are unable to read and comprehend English
9. Subjects are unable to provide informed consent
10. Other medical conditions for which these protocols are deemed inappropriate by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (A1C) | 1 year
  Change in HbA1c blood test
Blood pressure (systolic and diastolic blood pressure | 1 year
  Change in systolic and diastolic blood pressure reading
Lipids (LDLc, HDLc, cholesterol, and triglyceride) | 1 year
  Change in LDLc, HDLc, cholesterol, and triglyceride values

CONTACTS AND LOCATIONS:
Overall Officials: Janice Zgibor, RPh PhD, Principal Investigator — University of South Florida
Locations (1):
- University of Pittsburgh Medical Center Community Medicine Inc. (UPMC CMI) Primary Care Practices, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zgibor JC, Maloney MA, Malmi M Jr, Fabio A, Kuo S, Solano FX, Tilves D, Tu L, Davidson MB. Effectiveness of certified diabetes educators following pre-approved protocols to redesign diabetes care delivery in primary care: Results of the REMEDIES 4D trial. Contemp Clin Trials. 2018 Jan;64:201-209. doi: 10.1016/j.cct.2017.10.003. Epub 2017 Oct 6. PMID 28993287